CLINICAL TRIAL: NCT06695962
Title: Efficacy of Domperidone (a Prokinetic Agent) on Time in Range in Digestively Asymptomatic Type I Diabetic Patients with Delayed Gastric Emptying
Brief Title: Efficacy of Domperidone (a Prokinetic Agent) on Time in Range in Digestively Asymptomatic Type I Diabetic Patients with Delayed Gastric Emptying (Gastro-TIR)
Acronym: Gastro-TIR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/0380/HP
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetic
MeSH Terms: interventions — Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Domperidone then placebo (Experimental): Domperidone 10 mg, 3/days during 28 days, - wash-out (21 days) then placebo 3/days during 28 days
  Interventions: Drug: Domperidone 10mg; Drug: Placebo; Diagnostic Test: gastric emptying test
- Placebo then Domperidone (Experimental): Placebo 3/days during 28 days - wash-out (21 days) - then Domperidone 10 mg, 3/days during 28 days
  Interventions: Drug: Domperidone 10mg; Drug: Placebo; Diagnostic Test: gastric emptying test

INTERVENTIONS:
Drug: Domperidone 10mg — 30 mg per day for 21 days
Drug: Placebo — 3 per day for 21 days
Diagnostic Test: gastric emptying test — gastric emptying test

SUMMARY:
Patients living with type 1 diabetes PwT1D) still have trouble controlling their blood sugar, even with the latest treatments. PwT1D may have slow stomach emptying influencing blood glucose level. Treating this is an important goal. A recent study found that 30% of PwT1D had a slower gastric emptying rate, even though they had no other complications and were not experiencing any digestive issues. Slowing of gastric emptying is linked to gastric hypoglycaemia, which is a life-threatening condition that can affect quality of life, and to higher blood sugar level after eating. This can last throughout the night. Prokinetic treatments for the stomach are good for diabetic patients with slow digestion. They help with stomach pain and, to a lesser extent, with hypoglycemia. However, there is no data on the benefits of such treatments in patients with no digestive symptoms, on glycaemic control as defined by continuous glucose monitoring data. In fact, this may be more relevant than HbA1c in patients with alternating hypo- and/or hyperglycaemia.

We think that a prokinetic agent like domperidone could improve glycaemic control in PwT1D with slow gastric emptying and glycaemic imbalance.

This study tests how domperidone affects blood sugar levels in PwT1D. Patients will be administrated domperidone or a placebo for 28 days. We will see how long T1D patients spend within their blood sugar target range over 14 days using a continuous glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years and <75 years
* Known type 1 diabetic patients for > 5 years treated with multi-injection insulin regimen or insulin pump with continuous interstitial glucose recording device (CGM)
* Type 1 diabetic patients with glycemic target TIR (70-180 mg/dL) < 60% and/or CV > 40% and/or early postprandial hypoglycemia
* Patient with few symptoms of gastroparesis based on GCSI score ≤ 2
* Person who has read and understood the information letter and signed the consent form
* Person affiliated to a social security scheme
* A woman of childbearing potential (a woman is considered to be of childbearing potential fertile, after menarche and until she reaches menopause, unless she has reached the menopausal, unless she is definitively sterile)with at least effective contraception (i.e. at least: oral progestin-only hormonal contraception for which ovulation inhibition is not the primary mode of action, male or female condom with or without spermicide, cap, diaphragm or sponge with spermicide). for at least 1 month and a negative urine B-HCG pregnancy test at inclusion
* Surgically sterile women (hysterectomy, bilateral salpingectomy and bilateral oophorectomy)
* Menopausal women: The postmenopausal state is defined as the absence of menstrual periods for 12 months without any other medical cause. An elevated follicle-stimulating hormone (FSH) level in the post-menopausalinterval can be used to confirm a post-menopausal state in women not using hormonal contraception or hormone replacement therapy. However, in the absence of 12 months' amenorrhea, a single FSH measurement is insufficient

Exclusion Criteria:

* Type 2 diabetic patients
* Patients with CGM<70%
* Type 1 diabetic patients with glycemic target TIR (70-180 mg/dL) < 40%
* Patients with renal insufficiency (GFR<60 ml/min according to CKD-EPI formula),
* Patients with contraindications to DOMPERIDONE ARROW 10 mg film-coated tablet:

  * Hypersensitivity to the active substance or to one of the excipients
  * Pituitary prolactin tumor (prolactinoma)
  * Underlying heart disease such as congestive heart failure (NYHA stage ≥2),
  * Kalemia less than 3.7 mmol/L or greater than 5.5 mmol/L,
  * Magnesemia less than 0.7 mmol/L
  * Hepatic impairment (TGO, TGP, GGT>2N, TP<70% (unless on anticoagulant))
  * Known prolongation of cardiac conduction intervals, notably the QTc interval (QTc greater than 440 ms for men and greater than 460 ms for women)
  * Use of drugs that prolong the QTc interval (class IA antiarrhythmics (e.g. disopyramide, hydroquinidine, quinidine) and class III antiarrhythmics (e.g. amiodarone, dofetilide, dronedarone, ibutilide, sotalol), certain antipsychotics (e.g. haloperidol, pimozide, sertindole), certain antidepressants (e.g. citalopram, escitalopram), certain antibiotics (e.g. erythromycin, levifloxacin, moxifloxacin, spiramycin), certain antifungals (e.g. pentamidine, fluconazole), certain antimalarial drugs (in particular halofantrine, lumefantrine), certain digestive drugs (e.g. cisapride, dolasetron, prucalopride), certain antihistamines (e.g. mequitazine, mizolastine), certain anticancer drugs (e.g. toremifene, vandetanib, vincamine), certain other drugs (e.g. bepridil, diphemanil, methadone), apomorphine (unless the benefit of concomitant administration outweighs the risks, and only if the precautions recommended for concomitant administration are strictly observed).
  * Taking levodopa
  * Use of drugs that are potent or moderate inhibitors of CYP3A4: antiproteases, systemic azole antifungals, certain macrolide antibiotics (clarithromycin, telithromycin, azithromycin, roxithromycin, etc.), diltiazem, verapamil, etc.
  * Bradycardia (< 50 bpm)
  * Use ofmedication that induces bradycardia and hypokalemia
  * Presence of gastrointestinal bleeding, mechanicalobstruction or digestive perforation
  * Lactose contraindication: galactose intolerance, total lactase deficiency,glucose-galactose malabsorption syndrome
* Contraindication to gastric emptying test : - allergy to eggs, gluten, milk proteins, etc. - hepatic insufficiency - pulmonary diffusion disorders
* Contraindication to placebo (calcium content): hypercalcemia/hypercalciuria, known calcium lithiasis
* Pregnant, parturient or breast-feeding women, or those without proven effective contraception
* Person deprived of liberty by an administrative or judicial decision, or person under court protection, subguardianship or guardianship
* Person taking part in another trial / having taken part in another therapeutic trial (study involving a drug or medical device) which could interfere with the products or procedures being investigated within a period of 4 weeks prior to inclusion
* Any history of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or from giving informed consent
* Patients treated with a closed insulin loop

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentages of time spent within the TIR (Time In Range) glycemic target range (70-180 mg/dL) | 14 days after domperidone or placebo
  The difference of percentages of time spent within the TIR glycemic target range (70-180 mg/dL) recorded over 14 days under prokinetic treatment (domperidone) or placebo in T1D patients with gastroparesis and inadequate glycemic control

SECONDARY OUTCOMES:
Variation in glycemic control criteria : HbA1c assay | 14 days after domperidone of placebo
  Variation in HbA1c assay between domperidone and placebo (measurement of differences)
Variation in glycemic control criteria : Plasma fructosamine assay | 14 days after domperidone of placebo
  Variation in Plasma fructosamine assay between domperidone and placebo (measurement of differences)
Variation in glycemic control criteria : Insulin dose | 14 days after domperidone of placebo
  Variation in Insulin dose between domperidone and placebo (measurement of differences)
Safety | 105 days
  Number of AE and SAE

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Amiens, Amiens
  - CHU de CAEN, Caen
  - CH Dieppe, Dieppe
  - Centre Hospitalier Intercommunal Elbeuf, Louviers, Val de Reuil, Elbeuf
  - GH Le Havre, Le Havre
  - CHU de ROUEN, Rouen

IPD SHARING:
Plan to Share IPD: No